CLINICAL TRIAL: NCT04493255
Title: An Open-Label, Single-Dose Study to Determine the Metabolism and Elimination of [14C]E7090 in Healthy Male Subjects
Brief Title: A Study to Determine the Metabolism and Elimination of [14C]E7090 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E7090-E044-002; 2019-004957-10 (EudraCT Number)
Record Dates: First submitted 2020-07-15; First posted 2020-07-30 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy Participants; Phase 1; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E7090 (Experimental): Participants will receive 100 microcurie (μCi) of [14C]E7090 as a single 35 milligram (mg), capsule, orally on Day 1.
  Interventions: Drug: [14C]E7090

INTERVENTIONS:
Drug: [14C]E7090 — [14C]E7090, oral capsule.
  Other Names: E7090

SUMMARY:
The primary objective of this study is to determine the pharmacokinetics (PK) and excretion of E7090 and its metabolites in healthy male participants. Also, to assess the safety and tolerability of a single dose of E7090 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, healthy males, age greater than or equal to (>=) 35 years and less than or equal to (<=) 55 years old at the time of informed consent
2. Body Mass Index (BMI) of >=18 to <=32 kilogram per square meter (kg/m^2) at Screening
3. Provide written informed consent
4. Willing and able to comply with all aspects of the protocol
5. History of a minimum of 1 bowel movement per day

Exclusion Criteria:

1. Participant has participated in any clinical research study involving a radiolabeled investigational product within the 12 months prior to Day -1 (Baseline)
2. Participant has previously completed or withdrawn from this study or any other study investigating E7090 or previously received E7090
3. Participant has had exposure to significant diagnostic or therapeutic radiation (example: serial x-ray, computed tomography scan, barium meal) or has current employment in a job requiring radiation exposure monitoring within 12 months prior to Day -1
4. Participant has the following ocular disorders:

   1. Any previous history or current evidence of corneal disorder
   2. Any previous history or current evidence of active macular disorder (example: age-related macular degeneration, central serous chorioretinal disease)
5. Participants has a known history of clinically significant drug allergy at Screening or Baseline (Day -1)
6. Participants has a known history of food allergies or significant seasonal or perennial allergy
7. Participants is known to be human immunodeficiency virus positive at Screening
8. Participants has active viral hepatitis (B or C) as demonstrated by positive serology at Screening
9. Participant has a poor peripheral venous access, in the opinion of the investigator (or designee)
10. Participant received blood products within 2 months prior to Day -1, or donation of blood within 3 months prior to Screening, donation of plasma within 2 weeks prior to Screening, or donation of platelets from 6 weeks prior to Screening

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
feu: Percentage of Administered Radioactive Dose of [14C]E7090 Excreted in Urine | Up to Day 57
Cumulative feu: Cumulative Percentage of Administered Radioactive Dose of [14C]E7090 Excreted in Urine From 0 to tlast Hours | Up to Day 57
fef: Percentage of Administered Radioactive Dose of [14C]E7090 Excreted in Feces | Up to Day 57
Cumulative fef: Cumulative Percentage of Administered Radioactive Dose of [14C]E7090 Excreted in Feces From 0 to tlast Hours | Up to Day 57
feu+ef: Percentage of Administered Radioactive Dose excreted of [14C]E7090 in Combined Excreta (Urine and Feces) | Up to Day 57
Cumulative feu+ef: Cumulative Percentage of Administered Radioactive Dose excreted of [14C]E7090 in Combined Excreta (Urine and Feces) From 0 to tlast Hours | Up to Day 57
Cmax: Maximum Observed Plasma Concentration for [14C]E7090, E7090 and its Metabolites | Day 1: 0-672 hours post-dose
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for [14C]E7090, E7090 and its Metabolites | Day 1: 0-672 hours post-dose
AUC(0-24h): Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours Postdose for [14C]E7090, E7090 and its Metabolites | Day 1: 0-24 hours post-dose
AUC(0-t): Area Under the Concentration- time Curve From Time 0 to Time of Last Quantifiable Concentration for [14C]E7090, E7090 and its Metabolites | Day 1: 0-672 hours post-dose
AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for [14C]E7090, E7090 and its Metabolites | Day 1: 0-672 hours post-dose
T1/2: Terminal Elimination Phase Half-life for [14C]E7090, E7090 and its Metabolites | Day 1: 0-672 hours post-dose
CL/F: Apparent Total Body Clearance for E7090 | Day 1: 0-672 hours post-dose
Vd/F: Apparent Volume of Distribution for E7090 | Day 1: 0-672 hours post-dose
MPR AUC(0-inf): Metabolite to Parent Ratio For AUC(0-inf) of Metabolite to E7090, Corrected for Molecular Weights | Day 1: 0-672 hours post-dose

SECONDARY OUTCOMES:
Metabolic profile of E7090: Concentration of Metabolite of E7090 in Plasma, Urine, and Feces | Up to Day 57
  Blood, urine and feces samples will be collected and analyzed to estimate the concentration of metabolite of E7090 by Liquid Chromatography/ multiple-stage Mass Spectroscopy method.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Baseline up to Day 57
Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters Values | Baseline up to Day 29
Number of Participants With Clinically Significant Change From Baseline in Vital Signs Values | Baseline up to Day 29
Number of Participants With Clinically Significant Change From Baseline in 12 Lead Electrocardiogram (ECG) Findings | Baseline up to Day 29
Number of Participants With Any Suicidality Assessed Using Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline up to Day 29
  The C-SSRS is an interview-based rating scale to systematically assess any suicidality, any suicidal behavior, any suicidal ideation. Any suicidality: emergence of any suicidal ideation or suicidal behavior. Any suicidal behavior: when response is "yes" for any these questions- actual attempt to suicide, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation: when response is "yes" for any of these questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide. Number of participants with any suicidality will be reported for this outcome measure.
Number of Participants With Clinically Significant Change From Baseline in Ophthalmic Examinations | Baseline up to Day 29
  Ophthalmic examinations includes visual acuity, funduscopy, optical coherence tomography, and slit-lamp examination.
Number of Participants With Clinically Significant Change From Baseline in Physical Examinations | Baseline up to Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.